CLINICAL TRIAL: NCT04770506
Title: Prospective Interventional Study of Bone Mineral Density and Vascular Calcifications in the Population of Lithiasis Patients With Idiopathic Hypercalciuria
Brief Title: Bone Mineral Density and Vascular Calcifications in the Population of Lithiasis Patients With Idiopathic Hypercalciuria
Status: Completed | Type: Observational
Sponsor: Agnieszka Pozdzik (Other)
Responsible Party: Sponsor-Investigator, Agnieszka Pozdzik, Head of Dialysis Department, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Democles
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Hypercalciuria; Idiopathic
MeSH Terms: conditions — Hypercalciuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lithiasis patients: Lithiasis patients: diagnosis of recurrent NL confirmed by URO CT with presence of idiopathic hypercalciuria and metabolic workup available.
  Interventions: Other: Data extraction from medical files
- Control group: Control group: patients without NL matched for age and sex and who had a bone mineral densitometry or abdominal CT.
  Interventions: Other: Data extraction from medical files

INTERVENTIONS:
Other: Data extraction from medical files — Data extraction from medical files

SUMMARY:
In industrialized countries, it is estimated that around 10% of the population suffers from nephrolithiasis (NL). Numerous recent epidemiological studies report that the prevalence and incidence of NL continue to increase, with a prevalence that has nearly doubled over the past two decades. A patient who presented with a first episode of renal lithiasis has an estimated recurrence rate of nearly 50% at 5 years in adults. It is therefore wiser to consider NL as a chronic pathology and not as a simple isolated attack of painful crisis. NL therefore represents a real public health problem with a significant impact on the quality of life of patients, with considerable socio-economic repercussions.

In clinical practice, calcium lithiasis is the most common and occurs in 90% of cases.The stones mainly consist of calcium oxalate (whewellite, weddellite) but also calcium phosphate (carbapatite, brushite).

One of the risk factors for calcium lithiasis is the over-saturation of urine with calcium, which can lead to crystal formation.

The most common metabolic abnormality found in patients with NL is hypercalciuria.It is defined as an increased excretion of urinary calcium.We can first distinguish hypercalciuria secondary to another pathology such as primary hyperparathyroidism, sarcoidosis, distal tubular acidosis, hypervitaminosis D, immobilization... from idiopathic hypercalciuria (HI), at the origin of so-called primary calcium lithiasis.HI is estimated to affect 30-60% of adults with NL.

Idiopathic hypercalciuria is associated with low bone mineral density. Patients with NL have significantly lower T-score values in the vertebrae, hips, and femoral necks.Patients with NL have an increased risk of fractures and are 4 times more likely to develop osteoporosis. It is currently proposed that idiopathic hypercalciuria may be the cause of the decrease in bone mineral density in lithiasis patients.This bone demineralization appears to be associated with an increase in vascular calcifications.These, like NL, are believed to be linked to extra-osia calcium deposits.There is an inverse relationship between bone mineral density and arterial wall thickness (partly due to vascular calcifications) suggesting a relationship between arteriosclerosis and osteoporosis. This relationship would be much more pronounced in lithiasis women. In addition, several observations report an increase in cardiovascular morbidity in people with NL.

NL should therefore be seen as a systemic disease and is also associated with several pathologies such as: metabolic syndrome, arterial hypertension, diabetes and cardiovascular diseases.

To the knowledge of the investigators, no statistical data concerning the prevalence of vascular calcifications and bone demineralization in the population of lithiasis patients in Belgium has been published to date.

In this context, the aim of this study is to assess the prevalence of vascular calcifications (early state of arteriosclerosis) as well as the bone mineral density in the lithiasis population followed at the Brugmann University Hospital and with idiopathic hypercalciuria.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of recurrent NL confirmed by URO CT with presence of idiopathic hypercalciuria and metabolic workup available.

Exclusion Criteria:

People with stones other than calcium (uric acid, cysteine, infectious stones, indinavir stones, primary hyperoxaluria) or with secondary hypercalciuria (primary hyperparathyroidism, sarcoidosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of recurrent NL confirmed by URO CT with presence of idiopathic hypercalciuria and metabolic workup available.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-01-12 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
T-score | 5 minutes
  The T score is an indicator of bone mass provided by the dual energy x-ray absorptiometry (DXA) technique. The results are classified into four levels. Level 1: normal bone mass, level 2: osteopenia, level 3: osteoporosis, level 4: severe osteoporosis.
Aortic calcification index (ACI) | 5 minutes
  Estimations of aortic calcification are performed by abdominal computed tomography. ACI (%) = (total calcification score in all slices) / 12 (number of segments in each slice) x 10 (number of slices) x 100.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No